CLINICAL TRIAL: NCT07128381
Title: Phase I/II Clinical Trial of Axatilimab, a CSF1R Monoclonal Antibody, in Combination With Ruxolitinib as Therapy for Patients With Myelofibrosis (MF) and Chronic Myelomonocytic Leukemia (CMML)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0621; NCI-2025-05876 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis (MF); Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic | interventions — axatilimab; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy or Combination: Treatment with Axatilimab +/- Ruxolitinib IV Q4W (Experimental): Participants will self-administered approximately 12 hours apart without regard to food
  Interventions: Drug: Axatilimab (SNDX-6352); Drug: Ruxolitinib

INTERVENTIONS:
Drug: Axatilimab (SNDX-6352) — Taken orally
Drug: Ruxolitinib — Taken orally

SUMMARY:
* To find the recommended dose of axatilimab given alone and in combination with ruxolitinib in patients with MF and CMML.
* To learn if axatilimab given in combination with ruxolitinib can help to control MF and CMML.

DETAILED DESCRIPTION:
Primary Objectives:

* Phase 1 dose escalation: to determine safety, tolerability and Maximum Tolerated Dose (MTD) and efficacy of axatilimab alone and in combination with ruxolitinib for patients with MF and CMML
* Phase 2 dose expansion: to determine the overall response rate (ORR) of axatilimab and ruxolitinib in patients with MF and CMML.
* Incidence of AEs, MTD and changes in clinical laboratory values.
* Measures of efficacy in CMML: overall response rate (ORR) defined as sum of CR + complete cytogenetic remission + partial remission + marrow response + clinical benefit according to the IWG 2015 MDS/MPN response criteria37.
* Measures of efficacy in MF: objective response which is defined as CR (complete remission) + PR (partial remission) + CI (clinical improvement) after 6 cycles of treatment. It will be categorized according to the International Working Group (IWG) consensus criteria for myelofibrosis26

Secondary Objectives:

CMML:

* To determine other efficacy outcomes such as duration of response, leukemia-free survival (LFS), progression-free survival (PFS) and overall survival (OS).
* To evaluate symptom burden improvement assessed by Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF TSS).
* To evaluate changes in clonal composition and VAF of identified mutations with therapy
* To measure changes in cytokine profile and monocyte populations in peripheral blood and bone marrow.

MF:

* To explore time to response and duration of response
* To explore changes in bone marrow fibrosis
* To evaluate symptom burden improvement assessed by Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF TSS) (Appendix 1).
* To explore changes in dynamic of cytogenetics and molecular mutations: JAK2V617F, CALR, MPL (or other relevant molecular markers) in terms of allele burden or changes in cytogenetic abnormalities
* To measure changes in serum and bone marrow cytokine profile pre- and post-therapy

ELIGIBILITY:
Inclusion Criteria:

* Age .18 years as MF and CMML are very rare diseases in the pediatric population.
* Diagnosis of MF by WHO or ICC and:

  1. Phase 1 dose escalation (Cohort A and B): at least 1 prior therapy for MF or with suboptimal response after at least 3 months of therapy with a JAK inhibitor.
  2. Phase 2 dose expansion:

  i. Relapsed cohort (Cohort C): Patients with at least 1 prior MF therapy. or ii. JAKi-naive cohort (Cohort D): patients with newly diagnosed and treatment naive MF with intermediate .1 risk by DIPSS-plus (Appendix 2)
* Diagnosis of CMML refractory to treatment with hydroxyurea (for patients with proliferative CMML defined as WBC.13x109/L) or at least 4 cycles of treatment with hypomethylating agent, with relapse/progression after any number of cycles of hypomethylating agent therapy or who are intolerant of treatment with either therapy. Patients may have received prior therapy with other investigational agents or cytotoxic regimens.
* ECOG performance status ≤2
* Adequate hepatic function with total bilirubin </=3 x ULN, AST or A LT </= 3xULN unless related to disease involvement.
* Serum creatinine clearance >30mL/min and no end/stage renal disease (using Cockcroft-Gault).
* Prior hydroxyurea for control of leukocytosis or use of hematopoietic growth factors (eg, G-CSF, GM-CSF, procrit, aranesp, thrombopoietin) is allowed at any time prior to cycle 1 day 1 of therapy.
* Patient (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study. Non-English speaking patients may be consented.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
  * Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.
  * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who are currently receiving treatment for a malignancy (not including basal cell carcinoma, nonmelanoma skin cancer, cervical carcinoma in situ, early stage breast cancer or localized prostate cancer treated with hormone therapy). Patients with history of other cancers should be free of disease for at least 2 years prior to the Screening Visit or not requiring active treatment at the time of enrollment.
* Patients who are receiving any other investigational agents or with prior CSF1-R inhibitor therapy.
* Active, uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been initiated and, at the time of screening, there is no evidence of infection worsening, such as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs, or radiographic findings attributable to infection.
* Patients with evidence of active or latent tuberculosis. Prior to enrollment, patients should be evaluated for tuberculosis risk factors, and those at higher risk should be tested for latent infection. Risk factors include, but are not limited to, prior residence in or travel to countries with a high prevalence of tuberculosis, close contact with a person with active tuberculosis, and a history of active or latent tuberculosis where an adequate course of treatment cannot be confirmed.
* Patients who have a known malabsorption syndrome or other condition that may impair absorption of study medication (e.g., gastrectomy).
* History of acute or chronic pancreatitis.
* Active symptomatic myositis.
* Platelet count <50x109/L prior to enrollment and treatment initiation (for ruxolitinib combination cohorts only) except if related to either treatment for MF or CMML or treatment with cytotoxic therapy for any other reason.
* Pregnant women are excluded from this study because axatilimab and ruxolitinib are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated on study. These potential risks may also apply to other agents used in this study.
* Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], doublebarrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study.
* Female patients with reproductive potential who do not have a negative urine or blood betahuman chorionic gonadotropin (beta HCG) pregnancy test at screening.
* Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy within 7 days of therapy initiation.
* Patients with history of chronic hepatitis B or C, irrespective of surface antigen or viral load detection given risk of viral reactivation with JAK inhibitor therapy.
* Patients with history of HIV given risk of JAK inhibitor-related immune-suppression.
* New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <50 by echocardiogram or multigated acquisition (MUGA) scan.
* History of myocardial infarction or thromboembolic disease within the last 6 months or unstable/uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2033-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pemmaraju, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org